CLINICAL TRIAL: NCT01882530
Title: Prospective, Controlled Versus Placebo, Randomized, Double-blind Study, Evaluating the Value of Non-opioid Analgesic Combination (Based on Paracetamol, Nefopam, Ketoprofen) for Postoperative Analgesia.
Brief Title: Non-opioid Analgesic Combination With Morphine for Postoperative Analgesia.
Acronym: OCTOPUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Practice on postoperative pain management changed
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 130505A-32
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Post Operative Analgesia
Keywords: Post operative analgesia ;; Paracetamol ;; Ketoprofen ;; Nefopam ;; Morphine
MeSH Terms: interventions — Acetaminophen; Nefopam; Ketoprofen; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Control group C: Placebo (Placebo Comparator): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Morphine
- Group P: Paracetamol (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Paracetamol; Drug: Morphine
- Group N: Nefopam (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Nefopam; Drug: Morphine
- Group K: Ketoprofen (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Ketoprofen; Drug: Morphine
- Group PN: paracetamol and nefopam (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Paracetamol; Drug: Nefopam; Drug: Morphine
- Group PK: paracetamol and ketoprofen (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Paracetamol; Drug: Ketoprofen; Drug: Morphine
- Group NK: nefopam and ketoprofen (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Nefopam; Drug: Ketoprofen; Drug: Morphine
- Group PNK: paracetamol, nefopam and ketoprofen (Experimental): All patients will receive treatment intraoperatively (IV) in 30 minutes, 60 minutes before the end of the intervention, then postoperatively every 6 hours for 48 hours.
  Interventions: Drug: Paracetamol; Drug: Nefopam; Drug: Ketoprofen; Drug: Morphine

INTERVENTIONS:
Drug: Paracetamol
  Arms: Group P: Paracetamol; Group PK: paracetamol and ketoprofen; Group PN: paracetamol and nefopam; Group PNK: paracetamol, nefopam and ketoprofen
Drug: Nefopam
  Arms: Group N: Nefopam; Group NK: nefopam and ketoprofen; Group PN: paracetamol and nefopam; Group PNK: paracetamol, nefopam and ketoprofen
Drug: Ketoprofen
  Arms: Group K: Ketoprofen; Group NK: nefopam and ketoprofen; Group PK: paracetamol and ketoprofen; Group PNK: paracetamol, nefopam and ketoprofen
Drug: Morphine
  Other Names: All patients will receive morphine postoperatively (titration, then PCA).

SUMMARY:
The combination of different analgesic drugs and/or analgesia techniques is part of the standard management of postoperative analgesia. The analysis of the literature reveals a lack of comparison of the associations of non-opioid analgesic (NOA) with morphine for postoperative analgesia.

The objectives of this study are :

* comparing the morphine sparing effect of different combination of 3 NOA (paracetamol, nefopam, ketoprofen) for postoperative analgesia.
* determining whether the morphine-sparing effect is associated with or without a reduction in the incidence of morphine side effects.
* evaluating the effects of NOA on postoperative hyperalgesia.

DETAILED DESCRIPTION:
Since the description of the concept of balanced analgesia in the early 90's, the combination of different analgesic drugs and/or analgesia techniques is part of the standard management of postoperative analgesia. A recent survey conducted in France by Fletcher et al. showed that patients often received one or more NOA associated with an opioid. The benefit and risk of the use of opioids associated with NOA were recently reassessed as part of a formal recommendation of experts and detailed in a recent review. The analysis of the literature reveals a lack of comparison of the combinations of NOA with morphine for postoperative analgesia. For example, paracetamol and morphine in combination does not always allow a significant morphine-sparing effect compared with morphine alone and does not reduce the incidence of morphine side effects. A number of definitive answers has therefore yet to be found: Does NOA -morphine association allow an effective morphine-sparing effect? Is there an interest in prescribing several NOAs in association? If yes, what are the most interesting combinations in terms of morphine-sparing effect and safety?

Another question concerns the effects of NOA on postoperative hyperalgesia. This hyperalgesia, which results from surgery-related inflammation, is increased by consumption of morphine and not only contributes to the overall experience of postoperative pain but also to the chronicisation of postoperative pain. Since in clinical practice, hyperalgesia can be measured using specific tools (Von Frey filament type), our study will evaluate the anti-hyperalgesic effects of NOA on a subgroup of patients enrolled in the centers used to evaluate nociceptive thresholds.

The objectives of this study are :

* comparing the morphine sparing effect of different combination of 3 NOA (paracetamol, nefopam, ketoprofen) for postoperative analgesia.
* determining whether the morphine-sparing effect is associated with or without a reduction in the incidence of morphine side effects.
* evaluating the effects of NOA on postoperative hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years
* Receiving scheduled surgery requiring the use of a PCA to treat postoperative pain
* Patients with a written informed consent
* Patients with a written informed consent for the sub-study on hyperalgesia (patients in the centers concerned)
* Affiliate to a social security system

Exclusion Criteria:

* Allergy to morphine, paracetamol, nefopam or ketoprofen or to any of their excipients
* Absorption of morphine and / or NOA within 24 hours before surgery
* Absorption of methadone within 48 hours before surgery
* History of epilepsy
* Renal insufficiency (creatinin clearance <30 ml / min MDRD)
* Hepatic insufficiency
* Severe respiratory insufficiency
* Pregnancy or breastfeeding women
* History of seizures
* Symptomatic urethroprostatic disorders
* Angle-closure glaucoma
* Gastrointestinal, cerebrovascular or other evolving bleedings
* Active peptic ulcer or active gastritis
* Severe heart failure
* History of asthma triggered by taking ketoprofen or similar substances
* Disable adult person under guardianship
* Use of nitrous oxide during anesthesia protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2016-01-16 (Actual); Study Completion 2016-01-16 (Actual)

PRIMARY OUTCOMES:
Morphine consumption (mg), accumulated over 24 hours, measured by patient controlled analgesia (PCA). | Day 1

SECONDARY OUTCOMES:
Morphine consumption (mg) measured by patient controlled analgesia (PCA). | Day 2, day 3
Incidence of side effects associated with morphine: nausea, vomiting, sedation, urinary retention, pruritus. | Day 3
Area of hyperalgesia measured using a von Frey filament expressed in cm2, 48 hours after surgery (sub-study in 3 centers). | Day 2
Incidence of chronic pain assessed by a telephone questionnaire 3 months after surgery (sub-study in 3 centers). | Month 3
Global satisfaction (measured after treatment) | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: ERIC BELLISSANT, Study Chair — Rennes University Hospital
Locations (19):
- France (19):
  - Karine Nouette-Gaulain, Bordeaux
  - Marcel Chauvin, Boulogne
  - Hawa Keita-Meyer, Colombes
  - Dominique Fletcher, Garches
  - Pierre Albaladejo, Grenoble
  - Frédéric Aubrun, Lyon
  - Xavier Capdevila, Montpellier
  - Hervé Bouaziz, Nancy
  - Karim Asehnoune, Nantes
  - Marc Raucoules, Nice
  - Jacques Ripart, Nîmes
  - Anissa Belbachir, Paris
  - Emmanuel Marret, Paris
  - Jean-Xavier Mazoit, Paris
  - Marc Beaussier, Paris
  - Sébastien Bloc, Quincy-sous-Sénart
  - Jean-Marc Malinovsky, Reims
  - Marc Gentili, Saint-Grégoire
  - Vincent Minville, Toulouse

REFERENCES:
- [Derived] Beloeil H, Albaladejo P, Sion A, Durand M, Martinez V, Lasocki S, Futier E, Verzili D, Minville V, Fessenmeyer C, Belbachir A, Aubrun F, Renault A, Bellissant E; OCTOPUS group. Multicentre, prospective, double-blind, randomised controlled clinical trial comparing different non-opioid analgesic combinations with morphine for postoperative analgesia: the OCTOPUS study. Br J Anaesth. 2019 Jun;122(6):e98-e106. doi: 10.1016/j.bja.2018.10.058. Epub 2018 Dec 29. PMID 30915987